CLINICAL TRIAL: NCT01419132
Title: Effects of High Furosemide Doses Alone or With Hypertonic Saline on Troponin I Myocardial Release in Acute Decompensated Heart Failure: a Double Blind Study.
Brief Title: Troponin I Release After High Diuretic Doses
Acronym: Tra-HSS-Fur
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Gaspare Parrinello, Effects of High Furosemide Doses Alone or With Hypertonic Saline on Troponin I Myocardial Release in Acute Decompensated Heart Failure: a Double Blind Study., University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tra-HSS-Fur; 12/11 UNIPA-AOUP (Other: University of Palermo, Policlinico General Hospital)
Record Dates: First submitted 2011-08-15; First posted 2011-08-17 (Estimated); Last update posted 2011-11-01 (Estimated); Status verified 2011-10

CONDITIONS: ADHF
Keywords: furosemide; hypertonic saline solution; troponin I
MeSH Terms: interventions — Furosemide; Diuretics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High doses furosemide (Placebo Comparator): administration of furosemide alone
  Interventions: Drug: Furosemide
- HSS plus furosemide (Experimental): administration of hypertonic saline solution plus high doses of furosemide bid
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — 125-250 mg furosemide bid
  Other Names: diuretics
  Arms: HSS plus furosemide
Drug: Furosemide — 125-250 mf furosemide bid
  Other Names: diuretics
  Arms: High doses furosemide

SUMMARY:
High values of cardiac troponin (Ct) in acute heart failure (ADHF) identify patients (pts) at higher risk and worsened prognosis. A Ct increase during therapy indicates the need for more appropriate intervention, aimed at compensating cardiac disease and effectively minimizing myocardial wall stress and subsequent cytolysis. This study evaluated the effects of an intravenous high-dose of furosemide with or without small-volume hypertonic saline solution (HSS)on myocardial cytolysis in ADHF pts.

DETAILED DESCRIPTION:
After randomization, all patients included in the study underwent a complete physical examination, including a careful check of HF signs and symptoms, including BW measurement (in the morning before breakfast), supine and standing blood pressure (BP [the mean of 3 measurements]), and heart rate (HR). Fasting blood samples were drawn to determine the serum levels of Na, K, Cl, bicarbonate, albumin, uric acid, creatinine, urea, and glycemia on a daily basis during hospitalization, and this was continued until a clinically compensated state was obtained. The total daily output of urine was collected for measuring levels of creatinine clearance, urinary Na and K. A chest radiograph, electrocardiogram, and echocardiogram (prior to commencing therapy and again when discharged. In addition, BNP and TNI plasma levels will be evaluated for all patients on entry and at discharge. Each patient provided written informed consent prior to participating in the study.

In order to determine GFR, the MDRD formula (Modification of Diet in Renal Disease), involving 4 parameters, was deployed. It provides an estimate of GFR comparable or superior to other formulae, with the advantage of not requiring any anthropometric measurements. According to the MDRD, GFR can be estimated using the following formula: GFR (ml/min/1.73m2) = 175 x {[serum creatinine (mg / dL or μmol/L/88.4)] -1.154 x {age (years) }-0.203 x 0.742 if female and 1.21 if Afro-American. The estimating of GFR by means of the MDRD formula is a useful and valid tool with which to obtain an index of kidney function.

The echocardiography M / B mode color Doppler will be performed with a Vivid 7 echocardiograph, with patients in a supine position and slightly left lateral decubitus. The mitral flow and the time taken for the wave to return to baseline (DTE) were evaluated from the apical 4 room positions, placing the sample volume of pulsed Doppler at the peak of the valve leaflets during the opening. Subsequently, the speed of early diastolic movement (Ea) of mitral annulus, obtained from the 4 room projection placing the sample volume of pulsed tissue Doppler onto lateral corner of the annulus, was assessed as an index of left ventricular relaxation. By measuring the Ea wave and the E / Ea ratio, the PCWP was evaluated in a quantitative way according to the following formulae:

PCWP = 1.24 E / Ea + 1.91 for those in sinus rhythm PCWP = 0.821 E / Ea + 6.489 for those in atrial fibrillation. Calculating dp/dt. The calculating of dp/dt was performed by a spectral analysis of mitral regurgitation at CW Doppler. Two points were chosen on the mitral regurgitation curve for the correct calculation of echocardiographic dp / dt: A: speed 1 m / sec = 4 mm Hg; and B: speed 3 m / sec = 36 mm Hg. The pressure gradient between these two point was reported to be 32 mmHg (A - B = 36 - 4 = 32). dP/dT was calculated by dividing the pressure gradient between the two points for the temporal distance between them: dP / dT = 32mmHg / T msec.

Bioelectrical impedance variables will be detected with an impedance plethysmograph using a previously-described methodology (18). This emitted an alternating sinusoidal electric current of 800 mA and an operating single frequency of 50 kHz; it which was calibrated each morning using a standard resistor supplied by the manufacturer. BIA is a method for detecting whole-body fluid overload and pulmonary congestion, based on the theory that the accumulation of whole-body or intrathoracic fluid will conduct an electrical current passing across the body or trunk more easily, leading to a decrease in whole-body or pulmonary bioimpedance. Bioimpedance is a combination of resistance (Rz) (ie, the opposition of an alternating current flowing through intra- and extra-cellular ionic solutions) and reactance (Xc) (ie, the capacitative component of tissue interfaces, cell membranes, and organelles). As previous described, in standard whole-body tetrapolar BIA, sensing electrodes were placed on: the dorsum of the wrist, a line between the radial and ulnar styloid processes, the dorsum of the ipsilateral foot, and on a line between the medial and lateral malleoli. Source electrodes were placed to overlie the head of the third metacarpal on the dorsum of the hand and the third metatarsal on the dorsum of the foot, on the same side as the sensing electrodes. The measurements will be performed on the right side of the body with the patients in a semi-orthopneic or supine position. According to the RzXc graph method of the BIA vector, the impedance measurement will be standardized according to the height (H) of the subject, expressing both Rz/H and Xc/H in ohm/meters, to establish the hydration state. Bioelectrical impedance measurements will be assessed twice by the same experienced operator and paired measurements for each patient were used in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* signs/symptoms of heart failure;
* New York Heart Association (NYHA) functional Class III or IV on admission due to an exacerbation of symptoms with at least 1 class deterioration;
* evidence of systolic dysfunction on echocardiographic examination on admission (EF<45%);
* BNP levels on admission > 100pg/mL

Exclusion Criteria:

* NYHA class < III on admission or without a NYHA class improvement on discharge;
* acute coronary syndrome,
* pulmonary thromboembolism,
* cardiac tamponade,
* pericarditis,
* renal insufficiency (serum creatinine <2,5 mg/dL, BUN <60 mg/dL) or those on dialysis;
* chronic liver disease,
* pleuro-pneumonia,
* blood and autoimmune diseases,
* concomitant other important co-morbidity,
* cerebral vascular disease,
* dementia,
* cancer,
* uncompensated diabetes,
* took non-steroid anti-inflammatory drugs (NSAID)
* declining to provide informed consent,
* patients requiring pacemaker implantation and those with issues of excessive alcohol consumption

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
troponin I plasma levels (pg/ml) | participants will be followed for the duration of hospital stay, an expected average of 1 weeks
  troponin I will be evaluated at entry and at dicharge

CONTACTS AND LOCATIONS:
Overall Officials: Parrinello Gaspare, MD, Study Chair — University of Palermo
Locations (3):
- Italy (3):
  - Department of Internal and Specialty Medicine, Palermo, Palermo
  - Gaspare PArrinello, Palermo, Palermo
  - GF Ingrasasia Hospital, Palermo, Palermo

REFERENCES:
- [Result] Kociol RD, Pang PS, Gheorghiade M, Fonarow GC, O'Connor CM, Felker GM. Troponin elevation in heart failure prevalence, mechanisms, and clinical implications. J Am Coll Cardiol. 2010 Sep 28;56(14):1071-8. doi: 10.1016/j.jacc.2010.06.016. PMID 20863950
- [Result] Parrinello G, Paterna S, Di Pasquale P, Torres D, Mezzero M, Cardillo M, Fasullo S, La Rocca G, Licata G. Changes in estimating echocardiography pulmonary capillary wedge pressure after hypersaline plus furosemide versus furosemide alone in decompensated heart failure. J Card Fail. 2011 Apr;17(4):331-9. doi: 10.1016/j.cardfail.2010.11.003. Epub 2010 Dec 24. PMID 21440872
- [Derived] Parrinello G, Di Pasquale P, Torres D, Cardillo M, Schimmenti C, Lupo U, Iatrino R, Petrantoni R, Montaina C, Giambanco S, Paterna S. Troponin I release after intravenous treatment with high furosemide doses plus hypertonic saline solution in decompensated heart failure trial (Tra-HSS-Fur). Am Heart J. 2012 Sep;164(3):351-7. doi: 10.1016/j.ahj.2012.05.025. Epub 2012 Aug 17. PMID 22980301